CLINICAL TRIAL: NCT06252610
Title: PET/MRI Evaluation in Patients With Primary Sclerosing Cholangitis Using Intercellular Matrix Radiopharmaceuticals
Brief Title: PET/MRI of Primary Sclerosing Cholangitis
Status: Not yet recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Onofrio A. Catalano, MD, PhD, MD, Ph.D, Massachusetts General Hospital
Other Study IDs: 2022P002225
Record Dates: First submitted 2024-02-02; First posted 2024-02-09 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: PSC
Keywords: PSC; [18F]-FAPI-74; [68Ga]CBP8-PET; PET/MR; Fibrosis
MeSH Terms: conditions — Fibrosis | interventions — Contrast Media; Magnetic Resonance Spectroscopy; Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PSC: Population will be consecutive patients with PSC, who will be referred to us by the MGB-affiliated hepatologists.
  Interventions: Drug: Radiotracer Injection; Drug: Contrast Media, Magnetic Resonance; Diagnostic Test: Imaging

INTERVENTIONS:
Drug: Radiotracer Injection — An intravenous catheter will be placed in an arm or hand vein for injection of [68Ga]CBP8;
  * 6-10 mCi of [68Ga]CBP8 or 5-9 mCi of FAPI will be injected into the Biograph mMR system. The injected dose and the time of injection will be recorded;
  * The catheter will be flushed with 0.9% saline solution;
  * The subjects will then be positioned on the scanner table; support devices under the back or legs will be used to enable the patient to maintain his/her position throughout the scan comfortably.
Drug: Contrast Media, Magnetic Resonance — The same intravenous catheter used to inject the radiotracer will be used to inject the hepatospecific gadolinium contrast agent Eovist (Bayer, Whippany, NJ);
  * After being positioned on the PET/MRI table, the nuclear medicine technologist will connect the patient to the MRI-safe power injector;
  * The catheter will be flushed before and after injection with 0.9% saline solution;
  * About halfway through the imaging session, the study staff will inform the patient that they are going to be administering the contrast agent and what sensations they should and should not expect;
  * The contrast will then be injected.
Diagnostic Test: Imaging — MRI and PET scanner to be used:
  3.0 T Laboratory (Bay 7) Siemens Biograph mMR.
  Magnetic resonance images of the abdomen will be acquired using the Martinos Center's combined 3 Tesla PET/MRI scanner. The image quality on these 3 Tesla devices will be very high, equivalent to or better than any other standard clinical MRI system. PET images of the target body site will be acquired When necessary, the data acquisition will be started shortly before radiotracer injection; Coincidence event data will be acquired and stored in list mode or compressed (i.e., sinogram space) format. Subjects will be asked to lie still for the duration of the study. The entire imaging session will last up to 120 minutes

SUMMARY:
This study aims to use positron emission tomography (PET)/magnetic resonance imaging (MRI) to diagnose and quantify PSC-related biliary tract fibrosis and to improve upon the currently available non-invasive diagnostic capabilities by investigating the ability of combined PET/MRI to detect and quantify fibrosis using a novel collagen-binding radiotracer. Specifically, the investigators will be comparing [68Ga]CBP8- and [18F]-FAPI-74 PET/MRI to a liver transient elastography scan in the diagnosis of biliary tree fibrosis.

DETAILED DESCRIPTION:
Imaging in the form of cholangiography plays an essential role in diagnosing and managing PSC. In the past decade, magnetic resonance cholangiopancreatography (MRCP) has become preferred over endoscopic retrograde cholangiopancreatography (ERCP) for the diagnosis of PSC because it is non-invasive, thereby safer, and cheaper than ERCP. MRCP's sensitivity and specificity for diagnosing PSC are high, 86% and 94%, respectively. However, to quantify liver fibrosis, MRCP is only accurate in more advanced stages of the disease. Intrahepatic biliary stricture severity was a poor discriminator between the different grades of liver fibrosis measured on magnetic resonance elastography and the different risk strata according to the Mayo Risk Score and The Amsterdam-Oxford prognostic index (AOPI). Other non-invasive diagnostic tests, such as transient elastography, lack full-organ evaluation and may be subject to variation between measurements, despite being the current gold standard for non-invasive fibrosis quantification.

This study aims to use [68Ga]CBP8- or [18F]FAPI PET/MRI to diagnose and quantify PSC-related biliary tract fibrosis. The novel radiopharmaceutical collagen-binding probe 8 labeled with Gallium-68 selectively binds to collagen type I, the predominant extracellular protein in fibrosis. [68Ga]CBP8 has already been investigated in patients affected by pulmonary fibrosis with success. Fibroblast activation protein (FAP) is a type II transmembrane serine protease that is overexpressed in CAFs and, to a lesser extent, in benign processes. It is associated with extracellular matrix remodeling, for example, chronic inflammation, degenerative bone and spine disease, arthritis, and cardiac remodelling after myocardial infarction. Quinolone-based FAP inhibitors (FAPIs) constitute a class of molecules with high affinity to FAP deployed to assess many types of solid tumors and some benign pathologies. 68Ga-FAPIs and, to a lesser extent, 18F-FAPI are being extensively studied in oncologic and non-oncologic positron emission tomography/computed tomography (PET/CT) and, to a lesser extent, PET/MRI, both in Europe and Asia.

In this open-label, single-arm, single-center prospective study, the investigators will recruit 10 patients with known primary sclerosing cholangitis (PSC) who have previously undergone other modalities for the evaluation of hepatic fibrosis, such as liver biopsy and/or transient elastography (FibroScan) and/or MR liver elastography and/or US liver elastography.No healthy volunteers will be included. Patients will be referred to [68Ga]CBP8 or [18F]-FAPI-74 PET/MRI by their primary treating physicians (e.g., hepatologist). After a phone-call pre-screening, electronic medical records verification, and a screening visit, subjects will be imaged with [68Ga]CBP8 or [18F]-FAPI-74 PET/MRI. A blood draw might also be performed to measure serum biomarkers of liver fibrosis.

Transient liver elastography has a diagnostic accuracy ranging from 65% in the initial stages to 90% for severe fibrosis in the setting of PSC. There is no data regarding the use of [68Ga]CBP8 PET/MRI to diagnose or quantify fibrosis in PSC. Therefore, the investigators lack sufficient evidence to estimate power with a reasonable degree of certainty. By enrolling 10 patients for this initial pilot study in the evaluation of hepatic/biliary fibrosis with [68Ga]CBP8 PET/MRI, the investigators will be able to acquire enough data to determine the optimal sample size for a larger study. A paired McNemar's test will be used for hypothesis testing regarding differences in sensitivity, specificity, accuracy, negative predictive value, and positive predictive value between [68Ga]CBP8 PET/MRI and FibroScan. Moreover, the investigators will analyze quantitative features of PET (SUV) and obtain their correlation to the actual fibrosis as reported by the gold standard test. These will be performed using Spearman's correlation coefficient and regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Established clinical diagnosis of large duct PSC
* Participants receiving treatment for IBD are allowed if on a stable dose from screening and expected to remain stable for the duration of the study
* Serum AST and ALT concentration ≤ 8 times the upper limit of normal

Exclusion Criteria:

* Other causes of chronic liver disease, including secondary sclerosing cholangitis or viral, metabolic, or alcoholic liver disease, as assessed clinically
* Known or suspected overlapping clinical or histologic diagnosis of autoimmune hepatitis
* Subjects less than 18 years of age or greater than 85 years of age.
* Subjects with electrical implants, such as cardiac pacemakers or perfusion pumps.
* Subjects with ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, prosthetic heart valves that are not compatible with the gradient maps of our scanners, metal fragments, shrapnel, metallic tattoos anywhere on the body, tattoos near the eye, or steel implants ferromagnetic objects such as jewelry or metal clips in clothing.
* Subjects who anticipate being pregnant or breastfeeding (a negative STAT quantitative serum hCG pregnancy test is required on the day of the scan before the subject can participate).
* Subjects with claustrophobic reactions
* Subjects with more significant than average potential for cardiac arrest.
* Subjects with a history of major head trauma (i.e., multiple concussions, traumatic brain injury).
* Subjects with a history of bleeding disorders.
* Subjects whose research-related radiation exposure exceeds current Radiology Department guidelines (i.e., 50 mSv in the prior 12 months).
* Subjects unable to lie comfortably on a bed inside the PET/MRI bore as assessed by physical examination and medical history (e.g., back pain, arthritis).
* Subjects under the direct supervision of the principal investigator;
* Subjects with a body weight of > 300 lbs (operational weight limit of the PET/MRI table) or BMI >33 kg/m2 (the Athinoula A. Martinos Center standard procedure to avoid claustrophobia or mechanical impossibility of fitting the subject into the scanner bore, which is less than 60 cm wide).
* A history of acute or chronic severe renal insufficiency (glomerular filtration rate <30 mL/min/1.73m2
* Perioperative liver transplantation period.
* A history of systemic lupus, multiple myeloma, nephrogenic systemic fibrosis, or other comorbidities resulting in chronic kidney disease stage IV or higher

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In total, 10 subjects with PSC fulfilling the inclusion criteria will be recruited. All subjects recruited for the study will be able to withdraw from the study at any time. The patients will be referred to the study by their treating physicians to investigate liver or biliary tract fibrosis in the setting of PSC.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2026-05-10 (Estimated); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy in detection of fibrotic components in patients with PSC | (1-2 Months)
  To establish the diagnostic capabilities (sensitivity, specificity, accuracy) of PET/MRI using [68Ga]CBP8 or [18F]-FAPI-74 for detection of the fibrotic component in patients with PSC.
Quantification of fibrotic components in PSC | From date of PET/MRI examination to date of final histopathology result: (max. 1-2 Months)
  Quantification of fibrotic component in patients with PSC with [68Ga]CBP8- or [18F]-FAPI-74-PET/MT by using liver histology (when available) as the standard for comparison. If histology is unavailable, non-invasive tests (FibroScan, MRI Elastography, serum biomarkers) will be used.

SECONDARY OUTCOMES:
Correlation of PET parameters with clinical and imaging biomarkers/tests for fibrosis | 1-2 Months
  Compare fibrosis levels as measured by [68Ga]CBP8 or [18F]FAPI-74-PET/MRI to selected fibrosis plasma biomarkers, fibroscan, and derived scores.
Correlation of PET parameters with MRI parameters | 1-2 Months
  Compare fibrosis levels with gadoxetate contrast-enhanced and other MRI parameters (e.g., MRCP)

CONTACTS AND LOCATIONS:
Overall Officials: Onofrio Catalano, MD, Ph.D, Principal Investigator — Athinoula A. Martinos Center for Biomedical Imaging, Massachusetts General Hospital, Harvard Medical School
Locations (1):
- Athinoula A. Martinos Center for Biomedical Imaging, Massachusetts General Hospital, Harvard Medical School, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ludwig J. Surgical pathology of the syndrome of primary sclerosing cholangitis. Am J Surg Pathol. 1989;13 Suppl 1:43-9. PMID 2699167
- [Background] Lindor KD, Kowdley KV, Harrison ME; American College of Gastroenterology. ACG Clinical Guideline: Primary Sclerosing Cholangitis. Am J Gastroenterol. 2015 May;110(5):646-59; quiz 660. doi: 10.1038/ajg.2015.112. Epub 2015 Apr 14. PMID 25869391
- [Background] Dave M, Elmunzer BJ, Dwamena BA, Higgins PD. Primary sclerosing cholangitis: meta-analysis of diagnostic performance of MR cholangiopancreatography. Radiology. 2010 Aug;256(2):387-96. doi: 10.1148/radiol.10091953. PMID 20656832
- [Background] Tafur M, Cheung A, Menezes RJ, Feld J, Janssen H, Hirschfield GM, Jhaveri KS. Risk stratification in primary sclerosing cholangitis: comparison of biliary stricture severity on MRCP versus liver stiffness by MR elastography and vibration-controlled transient elastography. Eur Radiol. 2020 Jul;30(7):3735-3747. doi: 10.1007/s00330-020-06728-6. Epub 2020 Mar 4. PMID 32130494
- [Background] Vuppalanchi R, Sanyal AJ. Myths and mysteries about staging hepatic fibrosis by fibroscan. Clin Gastroenterol Hepatol. 2015 Apr;13(4):780-2. doi: 10.1016/j.cgh.2014.10.030. Epub 2014 Nov 5. No abstract available. PMID 25451885
- [Background] Montesi SB, Izquierdo-Garcia D, Desogere P, Abston E, Liang LL, Digumarthy S, Seethamraju R, Lanuti M, Caravan P, Catana C. Type I Collagen-targeted Positron Emission Tomography Imaging in Idiopathic Pulmonary Fibrosis: First-in-Human Studies. Am J Respir Crit Care Med. 2019 Jul 15;200(2):258-261. doi: 10.1164/rccm.201903-0503LE. No abstract available. PMID 31161770
- [Background] Catalano OA, Gee MS, Nicolai E, Selvaggi F, Pellino G, Cuocolo A, Luongo A, Catalano M, Rosen BR, Gervais D, Vangel MG, Soricelli A, Salvatore M. Evaluation of Quantitative PET/MR Enterography Biomarkers for Discrimination of Inflammatory Strictures from Fibrotic Strictures in Crohn Disease. Radiology. 2016 Mar;278(3):792-800. doi: 10.1148/radiol.2015150566. Epub 2015 Oct 5. PMID 26436860
- [Background] Catalano OA, Wu V, Mahmood U, Signore A, Vangel M, Soricelli A, Salvatore M, Gervais D, Rosen BR. Diagnostic performance of PET/MR in the evaluation of active inflammation in Crohn disease. Am J Nucl Med Mol Imaging. 2018 Feb 5;8(1):62-69. eCollection 2018. PMID 29531862
- [Background] Corpechot C, Gaouar F, El Naggar A, Kemgang A, Wendum D, Poupon R, Carrat F, Chazouilleres O. Baseline values and changes in liver stiffness measured by transient elastography are associated with severity of fibrosis and outcomes of patients with primary sclerosing cholangitis. Gastroenterology. 2014 Apr;146(4):970-9; quiz e15-6. doi: 10.1053/j.gastro.2013.12.030. Epub 2013 Dec 31. PMID 24389304
- [Background] Ehlken H, Wroblewski R, Corpechot C, Arrive L, Rieger T, Hartl J, Lezius S, Hubener P, Schulze K, Zenouzi R, Sebode M, Peiseler M, Denzer UW, Quaas A, Weiler-Normann C, Lohse AW, Chazouilleres O, Schramm C. Validation of Transient Elastography and Comparison with Spleen Length Measurement for Staging of Fibrosis and Clinical Prognosis in Primary Sclerosing Cholangitis. PLoS One. 2016 Oct 10;11(10):e0164224. doi: 10.1371/journal.pone.0164224. eCollection 2016. PMID 27723798
- [Background] Kratochwil C, Flechsig P, Lindner T, Abderrahim L, Altmann A, Mier W, Adeberg S, Rathke H, Rohrich M, Winter H, Plinkert PK, Marme F, Lang M, Kauczor HU, Jager D, Debus J, Haberkorn U, Giesel FL. 68Ga-FAPI PET/CT: Tracer Uptake in 28 Different Kinds of Cancer. J Nucl Med. 2019 Jun;60(6):801-805. doi: 10.2967/jnumed.119.227967. Epub 2019 Apr 6. PMID 30954939
- [Background] Altmann A, Haberkorn U, Siveke J. The Latest Developments in Imaging of Fibroblast Activation Protein. J Nucl Med. 2021 Feb;62(2):160-167. doi: 10.2967/jnumed.120.244806. Epub 2020 Oct 30. PMID 33127618
- [Background] Giesel FL, Adeberg S, Syed M, Lindner T, Jimenez-Franco LD, Mavriopoulou E, Staudinger F, Tonndorf-Martini E, Regnery S, Rieken S, El Shafie R, Rohrich M, Flechsig P, Kluge A, Altmann A, Debus J, Haberkorn U, Kratochwil C. FAPI-74 PET/CT Using Either 18F-AlF or Cold-Kit 68Ga Labeling: Biodistribution, Radiation Dosimetry, and Tumor Delineation in Lung Cancer Patients. J Nucl Med. 2021 Feb;62(2):201-207. doi: 10.2967/jnumed.120.245084. Epub 2020 Jun 26. PMID 32591493
- [Background] Sanchez-Crespo A. Comparison of Gallium-68 and Fluorine-18 imaging characteristics in positron emission tomography. Appl Radiat Isot. 2013 Jun;76:55-62. doi: 10.1016/j.apradiso.2012.06.034. Epub 2012 Aug 29. PMID 23063597